CLINICAL TRIAL: NCT05863806
Title: Comparison of Mulligan Mobilization and Transverse Friction Massage in Rotator Cuff Syndrome
Brief Title: Mulligan Mobilization vs Transverse Friction Massage in Rotator Cuff Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01494
Record Dates: First submitted 2023-05-04; First posted 2023-05-18 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Rotator Cuff Syndrome
Keywords: Mulligan mobilization; Transverse Friction Massage; Rotator cuff syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Single (Outcomes Assessor) no
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilzation (Experimental): MWM technique was carrying out in flexion, abduction, external and internal rotation directions. For this technique, participants were seated on a stretcher, and the physical therapist is standing opposite of the upper extremity that is treated. The internal hand of the physical therapist stabilizes participants' shoulder girdle and, with the thenar eminence of the other hand, performed a glide of the humeral head (this direction is the most suitable for treating such shoulder limitations).
  Participants were asked to flex the affected shoulder until the pain started while the physical therapist sustained the gliding force to the humeral head. The single session of MWM technique was last around 20 minutes, in 3 sets of 10 repetitions with a rest interval of 30 seconds between each sets.
  Interventions: Other: Mulligan Mobilzation
- Trasverse Friction Massage (Active Comparator): Transverse Friction Massage technique: Patients in the group B were receiving soft tissue massage (deep friction) is made to bend his/ her elbow to 90o and put forearm behind his/ her back, then lean back in half lying position. Thus arm is fixed in adduction and medial rotation. It was given in transverse direction for 10 - 12 minutes. Transverse friction massage was given twice a week with the gap of days for the first 3 week and then the repetition is increased to 3 to 4 times a week for the rest of duration.
  Interventions: Other: Trasverse Friction Massage

INTERVENTIONS:
Other: Mulligan Mobilzation — Participants were instructed that MWM, including shoulder movement, must be pain-free and should be immediately stopped if any pain is experienced during the treatment.
  The single session of MWM technique was last around 20 minutes, in 3 sets of 10 repetitions with a rest interval of 30 seconds between each sets.
  Arms: Mulligan Mobilzation
Other: Trasverse Friction Massage — Deep friction massage was given to rotator cuff tendon with the tip of index finger, which is reinforced by middle finger.
  It was given in transverse direction for 10 - 12 minutes. Transverse friction massage was Given twice a week with the gap of days for the first 3 week and then the repetition is increased to 3 to 4 times a week for the rest of duration.
  Arms: Trasverse Friction Massage

SUMMARY:
The aim of this research is to determine the Effects of Mulligan Mobilization and Transverse Friction Massage in Rotator Cuff Syndrome. Randomized clinical trials will be done at Northwest General Hospital, Peshawar. The sample size is 42. The subjects were divided in two groups, with 21 subjects in Group A and 21 in Group B. Study duration was of 6 months. Sampling technique applied was Non probability Purposive Sampling technique. Both males and females of aged 30-70 years with rotator cuff syndrome from grade (0-3) were included. Tools used in the study are Visual Analogue Scale (VAS), Goniometer, and DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire. Data was analyzed through SPSS 23.

DETAILED DESCRIPTION:
The rotator cuff syndrome is developed in the subacromial area by compression between the humerus and the coracoacromial arc of the long head of the subacromial bursa and the biceps tendon. The diagnosis of rotator cuff tendonitis and Bursitis is made on the basis of special tests and Examination. The rotator cuff tendons undergo degenerative alterations, the tendons between the humeral head and the coracoacromial arch are compressed and ischemia caused by impingement or elevated intramuscular pressure is all aspects of the physiopathology of RCS.

Highly exposed workers have frequently had RCS associated with biomechanical, psychological, and organizational aspects examined; this could affect generalizations to the entire working population who are exposed to varying degrees of work-related shoulder restrictions. The relationship between work structure and the risk of shoulder illnesses has been rarely investigated. Although various individual factors can raise the incidence of shoulder discomfort and RCS, biomechanical factors are significantly linked to both conditions (e.g., age).

Neer defined the syndrome as impingement of the rotator cuff tendons against the coracoacromial ligament, the anterior edge and undersurface of the anterior part of the acromion, and, often, the acromioclavicular joint. There is consensus that risk factors for shoulder MSDs are upper arm elevation and repeated or prolonged overhead activities in combination with other biomechanical variables (e.g., repetition, force). There is less proof that excessive repetition or rigid shoulder positions are separate risk factors.

The main focus in Rotator Cuff syndrome management is on promoting self-management, reducing pain, optimize function, and modifying the disease process and its effects. The primary treatment for Rotator Cuff syndrome conservatively is physiotherapy which includes strength training, modalities, resistance training and Kinesiotaping. Resistance exercise can reduce Shoulder pain severity and strength in participants with symptomatic Shoulder RCS. Exercise is suggested as the first-line intervention of choice with comparable outcomes but at a lower cost and with fewer associated hazards than surgical therapy in recent randomized controlled studies and systematic reviews. Despite this, there is little evidence that explains what an effective exercise programmed looks like in terms of the kind of exercise, the number of sets and repetitions, tolerable pain levels, duration, and environment.

Mulligan's mobilization with movement (MWM) is a joint mobilization treatment in which the patient actively engages in the uncomfortable action while receiving a manual accessory glide to one of the joint surfaces. Recent research found that in asymptomatic people applying MWM with a postero-lateral glide resulted in less muscular activity in the shoulder muscles . In accordance with Cyriax, Transverse friction massage leads in traumatic hyperemia, which boosts blood flow and lessens discomfort. It also stimulates mechanoreceptors and enhances tissue perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female are included
* Age between 30 to 70
* Partial rupture and suffering from rotator cuff syndrome(differentiation is made on type of tear from grade 0 to 3)
* No shoulder surgery
* Pain on palpation of rotator cuff muscle
* Two or more provocative tests should be positive which is used to rule out the tendonitis and bursitis.

Exclusion Criteria:

* Multiple shoulder pathologies.
* Bursitis
* Corticosteroid injections last month
* Orthopedic or cardiovascular problem
* Recent myocardial infarction or major shoulder trauma

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Disability of Arm, Shoulder and Hand Questionnaire | 6th week
  Change from baseline the DASH score at 3rd and 6th week. The DASH (Disabilities of the Arm, Shoulder and Hand) Outcome Measure is a 30-item, self-report questionnaire that measures physical function and symptoms in people with musculoskeletal disorders of the upper limb. Changes from the baseline, and then at 3rd and 6th week

SECONDARY OUTCOMES:
Change from baseline in Visual Analogue Scale | 6th week
  Change from baseline the Visual Analogue Scale score at 3rd and 6th week. A device used by physical therapists to measure joints' range of motion. During measurement fulcrum will be placed on shoulder joint parallel to sagittal axis for abduction and adduction, frontal axis for flexion and extension and to humeral longitudinal axis in 90o of abduction for internal and external rotations. Changes from the baseline, and then at 3rd and 6th week

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University; Asad Khan, MSPT*, Principal Investigator — Northwest General Hospital
Locations (1):
- Northwest General Hospital and Research Center, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No